CLINICAL TRIAL: NCT05325164
Title: Methadone for 'Adenocarcinopathic' Pain Treatment: Methadone vs. Morphine Vanguard RCT
Brief Title: Methadone for 'Adenocarcinopathic' Pain Treatment
Acronym: METHADOPT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial not started; change in Sponsor and Principal Investigator, trial to be registered again by new Sponsor/Investigator if it is started.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Bruyère Health Research Institute. (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 638423678
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Cancer Pain; Adenocarcinoma
Keywords: Cancer; Methadone; Morphine; Hydromorphone; Adenocarcinoma
MeSH Terms: conditions — Cancer Pain; Adenocarcinoma; Neoplasms | interventions — Methadone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methadone (Experimental): DESCRIPTION:
  Blinded methadone 1mg tablets PO
  --
  DOSAGE:
  A) For patients initially taking 0-30 mg MEDD:
  Starting dose: 0.5mg Q4H x 4 doses + 1.0mg QHS + 0.5mg Q2H PRN (max 4 doses)
  First increase: 1.0 mg Q4H x 4 doses + 2.0mg QHS + 0.5mg Q2H PRN (max 4 doses)
  Second increase: 1.5mg Q4H x 4 doses + 3.0mg QHS + 0.5mg Q2H PRN (max 4 doses)
  Third increase: 2.0mg Q4H x 4 doses + 4.0mg QHS + 1.0mg Q2H PRN (max 4 doses)
  Fourth increase: 2.5mg Q4H x 4 doses + 5.0mg QHS + 1.0mg Q2H PRN (max 4 doses)
  B) For patients initially taking 31-60 mg MEDD:
  Starting dose: 1.0mg Q4H x 4 doses + 2.0mg QHS + 0.5mg Q2H PRN (max 4 doses)
  First increase: 1.5mg Q4H x 4 doses + 3.0mg QHS + 1.0mg Q2H PRN (max 4 doses)
  Second increase: 2.0mg Q4H x 4 doses + 4.0mg QHS + 1.0mg Q2H PRN (max 4 doses)
  Third increase: 2.5mg Q4H x 4 doses + 5.0mg QHS + 1.5mg Q2H PRN (max 4 doses)
  Fourth increase: 3.0mg Q4H x 4 doses + 6.0mg QHS + 1.5mg Q2H PRN (max 4 doses)
  Interventions: Drug: Methadone
- Morphine (Active Comparator): DESCRIPTION:
  Blinded morphine 5mg tablets PO
  --
  DOSAGE:
  A) For patients initially taking 0-30 mg MEDD:
  Starting dose: 2.5mg Q4H x 4 doses + 5.0mg QHS + 2.5mg Q2H PRN (max 4 doses)
  First increase: 5.0 mg Q4H x 4 doses + 10.0mg QHS + 2.5mg Q2H PRN (max 4 doses)
  Second increase: 7.5mg Q4H x 4 doses + 15.0mg QHS + 2.5mg Q2H PRN (max 4 doses)
  Third increase: 10.0mg Q4H x 4 doses + 20.0mg QHS + 5.0mg Q2H PRN (max 4 doses)
  Fourth increase: 12.5mg Q4H x 4 doses + 25.0mg QHS + 5.0mg Q2H PRN (max 4 doses)
  B) For patients initially taking 31-60 mg MEDD:
  Starting dose: 5.0mg Q4H x 4 doses + 10.0mg QHS + 2.5mg Q2H PRN (max 4 doses)
  First increase: 7.5mg Q4H x 4 doses + 15.0mg QHS + 5.0mg Q2H PRN (max 4 doses)
  Second increase: 10.0mg Q4H x 4 doses + 20.0mg QHS + 5.0mg Q2H PRN (max 4 doses)
  Third increase: 12.5mg Q4H x 4 doses + 25.0mg QHS + 12.5mg Q2H PRN (max 4 doses)
  Fourth increase: 15.0mg Q4H x 4 doses + 30.0mg QHS + 12.5mg Q2H PRN (max 4 doses)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — Methadone
  Other Names: Dolophine; Methadose
  Arms: Methadone
Drug: Morphine — Morphine
  Other Names: MS Contin; Kadian
  Arms: Morphine

SUMMARY:
Methadone is an opioid that has been used for over 80 years to treat various types of pain, including cancer pain. Despite its increasing popularity as a co-analgesic and first-line treatment for cancer pain, there remain some outstanding questions regarding its use in treating cancer pain, such as its efficacy compared to other opioids and its appropriateness as a first-line treatment. The investigators will conduct a Vanguard Randomized Clinical Trial (RCT) to estimate the efficacy of methadone compared to morphine for the treatment of a newly defined type of cancer pain, which the investigators have termed 'adenocarcinopathic' pain (ACPP).

DETAILED DESCRIPTION:
Background:

Methadone is an opioid that has been used for over 80 years to treat various types of pain, including cancer pain. Its use as a co-analgesic and first-line treatment for cancer pain is becoming more widespread. Despite its increasing popularity, there remain some outstanding questions regarding its use in treating cancer pain, such as its efficacy compared to other opioids and its appropriateness as a first-line treatment.

Traditional classifications of cancer related chronic pain is classified as neuropathic and nociceptive (somatic or visceral). This classification is based on clinical descriptors as opposed to pathophysiologic mechanisms. The investigators propose a new mechanism, called 'adenocarcinopathic' pain (ACPP), which can be defined as pain caused by an adenocarcinoma that is in 'proximity' to or invading a nerve or nerve plexus. The suggested mechanism of ACPP is that the tumour excretes excess glutamate, which activates NMDA receptors on nearby sensory nerves, causing the pain sensation. As methadone is an NMDA antagonist (and mu receptor agonist), it becomes an interesting molecule for ACPP in comparison to other opioids (such as morphine) that are unable to suppress NMDA receptors.

Study Hypothesis:

Methadone will demonstrate superior efficacy to morphine for the treatment of ACPP, and physicians will demonstrate satisfactory confidence in its use.

Study Objectives:

1. Monitor safety and response to treatment
2. Evaluate the confidence of physicians

Study Design:

Participants will be randomized to receive either methadone or morphine. Patients will be observed for a period of 14 days, plus one physician follow-up after 28 days.

Sample Size & Study Population:

The investigators will aim to enrol n=40 patients total across all sites. Eligible outpatients are those for whom a strong opioid is being initiated or escalated for the treatment of ACPP.

Intervention:

For patients previously taking 0-30mg morphine equivalent daily dose (MEDD), starting dose is 0.5mg Q4H for methadone, 2.5mg for morphine. For those previously taking 31-60 mg MEDD, starting dose is 1.0mg Q4H for methadone, 5.0mg for morphine. Up to 4 breakthrough analgesia doses allowed per day. Dose escalations can be made at each patient encounter according to a standard dosing schedule.

Study Outcome Measures:

Using validated questionnaires, the patient's degree of pain control & relief, degree of satisfaction, global impression of change, and any side effects will be assessed. In addition, physicians will be asked to rate their confidence in treating each patient.

Expected Outcomes:

Positive results should provide justification to prolong the study to complete a phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Cancer type is adenocarcinoma;
* In the physician's opinion, mechanism of pain is most likely linked to an adenocarcinoma 'in proximity to' or invading a nerve or nerve plexus (i.e., 'adenocarcinopathic' pain; ACPP);
* Experiencing poorly controlled pain (defined as pain of 4 or higher on a 10-point visual analogue scale) despite the use of non-opioid analgesics or despite the regular use of up to 60 mg morphine equivalent daily dose (MEDD);
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2;
* Estimated prognosis of at least 3 months;
* Able to fill out questionnaires and understand procedures in English and/or French;
* Able to provide first person informed consent;
* Physician deems it appropriate to start the patient on the opioid.

Exclusion Criteria:

* Known QTc prolongation (QTc greater than 500ms, QRS less than 120ms) or known congenital QTc prolongation syndrome;
* Taking at least one medication that increases risk of Torsades de Pointes (TdP): cisapride, disopyramide, dofetilide, flecainide, procainamide, propafenone, quinidine, quinine, sotalol;
* History of opioid abuse or dependence using Edmonton Pain Classification;
* Has geographic difficulties with follow-up in person;
* Has any of the following comorbidities: documented class 3 or 4 New York Heart Association (NYHA) heart failure, myocardial infarction in the last 3 months, unstable angina, pericardial disease, oxygen dependent pulmonary diseases, Parkinson's disease, suspected or diagnosed dementia, bipolar disorder, poorly managed major depression (current or treated) or anxiety disorder;
* Taking medication known to have clinically significant interactions with the CYP450 enzyme: carbamazepine, efavirenz, phenobarbital, rifampicin, azole antifungals, antiretrovirals, grapefruit juice, clarithromycin, erythromycin;
* Diagnosed with Child-Pugh class B and/or C cirrhosis;
* Has hepatic insufficiency, defined as jaundice with irreversible hyperbilirubinemia of at least 34 micromol/L despite biliary tract stents (severity criteria in Child-Pugh-Turcotte score);
* Received radiation or any nerve block or plexus block on the same side as the pain in the past 14 days or PLANNED within the next 14 days;
* PLANNED prescription for daily co-analgesia with pregabalin, gabapentin, or dexamethasone during the next 14 days (not including dexamethasone with chemotherapy);
* Taking medication associated with major risk of serotonin syndrome (monoamine oxidase inhibitors; MAOIs): linezolid, moclobemide, rasagiline, selegiline;
* Taking medication known to be an opioid agonist, antagonist, or partial agonist: naltrexone, buprenorphine, tapentadol, tramadol;
* Other negative characteristic as per physician discretion (e.g., reduced renal function).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Pain control | 2 weeks
  Proportion of patients reporting pain of 3 or less on a 10-point scale

SECONDARY OUTCOMES:
Pain control | 1 week
  Proportion of patients reporting pain of 3 or less on a 10-point scale
Pain relief | 1 week
  Proportion of patients reporting at least 50% pain relief since start of treatment
Pain relief | 2 weeks
  Proportion of patients reporting at least 50% pain relief since start of treatment
Patient satisfaction | 1 week
  Proportion of patients who are satisfied (yes or no) with their current level of pain control
Patient satisfaction | 2 weeks
  Proportion of patients who are satisfied (yes or no) with their current level of pain control
Physician confidence | 2 weeks
  Proportion of patients for whom physicians felt confident in treating with methadone or morphine
Global change | 2 weeks
  Patient's global impression of change (PGIC)
Side effects | 2 weeks
  Proportion of patients who experienced or had worsening opioid side effects

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gagnon, MD MSc, Principal Investigator — Centre de recherche du CHU de Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruera E, Palmer JL, Bosnjak S, Rico MA, Moyano J, Sweeney C, Strasser F, Willey J, Bertolino M, Mathias C, Spruyt O, Fisch MJ. Methadone versus morphine as a first-line strong opioid for cancer pain: a randomized, double-blind study. J Clin Oncol. 2004 Jan 1;22(1):185-92. doi: 10.1200/JCO.2004.03.172. PMID 14701781
- [Background] Mercadante S, Bruera E. Methadone as a First-Line Opioid in Cancer Pain Management: A Systematic Review. J Pain Symptom Manage. 2018 Mar;55(3):998-1003. doi: 10.1016/j.jpainsymman.2017.10.017. Epub 2017 Nov 1. PMID 29101087
- [Background] Haumann J, Geurts JW, van Kuijk SM, Kremer B, Joosten EA, van den Beuken-van Everdingen MH. Methadone is superior to fentanyl in treating neuropathic pain in patients with head-and-neck cancer. Eur J Cancer. 2016 Sep;65:121-9. doi: 10.1016/j.ejca.2016.06.025. Epub 2016 Aug 3. PMID 27494037
- [Background] Leppert W, Zajaczkowska R, Wordliczek J, Dobrogowski J, Woron J, Krzakowski M. Pathophysiology and clinical characteristics of pain in most common locations in cancer patients. J Physiol Pharmacol. 2016 Dec;67(6):787-799. PMID 28195060
- [Background] Slosky LM, BassiriRad NM, Symons AM, Thompson M, Doyle T, Forte BL, Staatz WD, Bui L, Neumann WL, Mantyh PW, Salvemini D, Largent-Milnes TM, Vanderah TW. The cystine/glutamate antiporter system xc- drives breast tumor cell glutamate release and cancer-induced bone pain. Pain. 2016 Nov;157(11):2605-2616. doi: 10.1097/j.pain.0000000000000681. PMID 27482630
- [Background] Gagnon B, Almahrezi A, Schreier G. Methadone in the treatment of neuropathic pain. Pain Res Manag. 2003 Fall;8(3):149-54. doi: 10.1155/2003/236718. PMID 14657982